CLINICAL TRIAL: NCT06612931
Title: Comparison of Dual-lumen Catheter-guided Mini-forceps Biopsy and Brush Cytology with Vacuum Aspiration in Suspicious Biliary Strictures: a Multicenter, Randomized, Crossover Trial
Brief Title: Comparison of Dual-lumen Catheter-guided Mini-forceps Biopsy and Brush Cytology with Vacuum Aspiration in Suspicious Biliary Strictures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Xijing Hospital of Digestive Diseases (Other); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Baiwen Li, Director of the Gastrointestinal Endoscopy Center, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2022108
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography (ERCP); Miniforceps Biopsy; Biliary Strictures; Brush Cytology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CMB (Experimental): In ERCP procedures, catheter-guided mini-forceps biopsy (CMB) is performed before biliary brush cytology with vacuum aspiration (BCA).
  Interventions: Procedure: Dual-lumen catheter-guided mini-forceps biopsy is performed first
- BCA (Active Comparator): In ERCP procedures, biliary brush cytology with vacuum aspiration (BCA) is performed before dilation catheter-guided mini-forceps biopsy (CMB).
  Interventions: Procedure: Biliary brush cytology with vacuum aspiration is performed first

INTERVENTIONS:
Procedure: Dual-lumen catheter-guided mini-forceps biopsy is performed first — In ERCP procedures, catheter-guided mini-forceps biopsy is performed before biliary brush cytology.
  Arms: CMB
Procedure: Biliary brush cytology with vacuum aspiration is performed first — In ERCP procedures, biliary brush cytology with vacuum aspiration is performed before dilation catheter-guided mini-forceps biopsy.
  Arms: BCA

SUMMARY:
In this randomized crossover trial involving patients with indeterminate biliary strictures, we aimed to compare the diagnostic performance of the dual-lumen catheter-guided miniforceps biopsy (CMB) device with that of brush cytology under aspiration (BCA).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-88 years old.
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study.
* Biliary obstructive symptoms,or indeterminate biliary stricture suspected to be intrinsic based on prior imaging.

Exclusion Criteria:

* Any contraindications to ERCP.
* Severe cardiopulmonary disease or coagulopathy.
* Biliary strictures caused by extrinsic compression.
* Unwillingness or inability to provide consent.
* Pregnant or breastfeeding women.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy | 6 months
  The accuracy of dual-lumen catheter-guided miniforceps biopsy (CMB) and brush cytology with vacuum aspiration (BCA) in the diagnosis of biliary strictures.

SECONDARY OUTCOMES:
the diagnostic sensitivity | 6 months
  The diagnostic sensitivity of dual-lumen catheter-guided mini-forceps biopsy and brush cytology with vacuum aspiration to the suspicious biliary strictures.
The diagnostic specificity | 6 months
  The diagnostic specificity of dual-lumen catheter-guided mini-forceps biopsy and brush cytology with vacuum aspiration to the suspicious biliary strictures.
Severe adverse events rates | 6 months
  The incidence of adverse events, namely, post-ERCP pancreatitis, gastrointestinal perforation, and bleeding were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Baiwen Li, Ph.D., Principal Investigator — Department of Gastroenterology, Shanghai General Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Department of Gastroenterology, Shanghai General Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: Undecided